CLINICAL TRIAL: NCT00002471
Title: Phase II Trial of Intensive, Short-Course Combination Chemotherapy in the Treatment of Newly Diagnosed Patients With Poor-Risk Nonlymphoblastic Lymphoma and Acute B-Lymphoblastic Leukemia and in Patients With Recurrent Non-Hodgkin's Lymphoma
Brief Title: Combination Chemotherapy in Treating Patients With Acute B-Lymphoblastic Leukemia or Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Purpose: Treatment
Other Study IDs: 90-013; CDR0000076672 (Registry Identifier: PDQ (Physician Data Query)); NYU-97-9; NCI-V90-0104
Record Dates: First submitted 1999-11-01; First posted 2004-08-30 (Estimated); Last update posted 2013-06-20 (Estimated); Status verified 2013-06

CONDITIONS: Leukemia; Lymphoma
Keywords: childhood Burkitt lymphoma; L3 childhood acute lymphoblastic leukemia; B-cell childhood acute lymphoblastic leukemia; L3 adult acute lymphoblastic leukemia; B-cell adult acute lymphoblastic leukemia; recurrent adult non-Hodgkin lymphoma; stage III adult diffuse large cell lymphoma; stage III adult immunoblastic large cell lymphoma; stage III adult Burkitt lymphoma; stage IV grade 3 follicular lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult Burkitt lymphoma; recurrent grade 3 follicular lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult Burkitt lymphoma; stage III childhood small noncleaved cell lymphoma; stage IV childhood small noncleaved cell lymphoma; stage IV childhood large cell lymphoma; recurrent childhood small noncleaved cell lymphoma; recurrent childhood large cell lymphoma
MeSH Terms: conditions — Leukemia; Lymphoma; Burkitt Lymphoma; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Lymphoma, Follicular; Dendritic Cell Sarcoma, Interdigitating | interventions — Asparaginase; Cyclophosphamide; Cytarabine; Daunorubicin; Dexamethasone; Etoposide; Leucovorin; Methotrexate; Methylprednisolone; Hydrocortisone; Thiotepa; Vincristine

INTERVENTIONS:
Drug: asparaginase
Drug: cyclophosphamide
Drug: cytarabine
Drug: daunorubicin hydrochloride
Drug: dexamethasone
Drug: etoposide
Drug: leucovorin calcium
Drug: methotrexate
Drug: methylprednisolone
Drug: therapeutic hydrocortisone
Drug: thiotepa
Drug: vincristine sulfate

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Combining more than one drug may kill more cancer cells.

PURPOSE: Phase II trial to study the effectiveness of combination chemotherapy in treating patients who have acute B-lymphoblastic leukemia or recurrent non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES: I. Improve the survival of children and adolescents with poor-risk nonlymphoblastic lymphoma and acute B-lymphoblastic leukemia using an intensive, short-course regimen of combination chemotherapy. II. Assess the toxicity of the regimen.

OUTLINE: Nonrandomized study. Induction: 7-Drug Combination Chemotherapy with Leucovorin Rescue plus Triple Intrathecal Therapy (TIT). Cyclophosphamide, CTX, NSC-26271; Thiotepa, TSPA, NSC-6396; Vincristine, VCR, NSC-67574; Daunorubicin, DNR, NSC-82151; Dexamethasone, DM, NSC-34521; Etoposide, VP-16, NSC-141540; Methotrexate, MTX, NSC-740; with Leucovorin calcium, Citrovorum Factor, CF, NSC-3590; plus TIT: IT MTX; IT Cytarabine, IT ARA-C, NSC-63878; IT Hydrocortisone, IT HC, NSC-10483. Consolidation: 6-Drug Combination Chemotherapy with Leucovorin Rescue plus TIT. ARA-C; VP-16; Asparaginase (E. coli), ASP, NSC-109229; MTX; VCR; Methylprednisolone, MePRDL, NSC-19987; with CF; plus TIT. Reinduction: 7-Drug Combination Chemotherapy with Leucovorin Rescue plus TIT. CTX; TSPA; VCR; DNR; DM; VP-16; MTX; with CF; plus TIT.

PROJECTED ACCRUAL: A maximum of 30 patients, accrued from 4 institutions, will be entered. If at any time more than 3 patients are not "event free", the trial will be terminated early, with patients considered event free if they enter remission, do not die as a result of treatment toxicity, and do not experience progression within 1 year from the start of therapy.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Newly diagnosed undifferentiated nonlymphoblastic non-Hodgkin's lymphoma (Burkitt's or non-Burkitt's) Newly diagnosed large cell lymphoma with CNS involvement Recurrent non-Hodgkin's lymphoma L-3 and B-cell leukemia included At least 1 of the following required: LDH at least 500 IU/liter (old method) or 2,000 IU/liter (new method) Bone marrow involvement (greater than 5% lymphoblasts) CNS involvement (lymphoblasts on CSF cytospin or intracranial mass on CT or MRI scan)

PATIENT CHARACTERISTICS: Age: Any age Performance status: Not specified Hematopoietic: Not specified Hepatic: Not specified Renal: Not specified

PRIOR CONCURRENT THERAPY: Prior therapy allowed for non-Hodgkin's lymphoma No prior therapy for all other diseases

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1990-02; Primary Completion 2003-01 (Actual); Study Completion 2003-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Norma Wollner, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (4):
- United States (4):
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Kaplan Cancer Center, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania

REFERENCES:
- [Background] Finlay JL, Wasserman R, Willoughby M, et al.: A pilot study of brief intensive chemotherapy for children with high-risk small non-cleaved cell lymphoma (SNCCL) and acute B-cell leukemmia (B-ALL). Med Pediatr Oncol 21(8): A-18, 535, 1993.